CLINICAL TRIAL: NCT04608331
Title: Impact of Dexmedetomidine Supplemented Analgesia on Sleep Quality in Patients at High-risk of Obstructive Sleep Apnea After Major Surgery: A Randomized, Double-blind, and Placebo-controlled Pilot Study
Brief Title: Dexmedetomidine Supplemented Analgesia in Patients at High-risk of Obstructive Sleep Apnea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-189
Record Dates: First submitted 2020-10-21; First posted 2020-10-29 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Obstructive Sleep Apnea; Analgesia; Dexmedetomidine; High-flow Nasal Cannula; Sleep Quality
Keywords: Obstructive Sleep Apnea; Analgesia; Dexmedetomidine; High-flow nasal cannula; Sleep quality
MeSH Terms: conditions — Sleep Apnea, Obstructive; Agnosia; Sleep Initiation and Maintenance Disorders | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Patient-controlled analgesia is established with morphine (0.5 mg/ml) and dexmedetomidine (1.25 microgram/ml) in a total volume of 160 ml. The pump is programmed to deliver 2-ml boluses at 6 to 8-minute lockout intervals with a background infusion rate at 1 ml/h. Patient-controlled analgesia is provided for at least 24 hours after surgery.
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): Patient-controlled analgesia is established with morphine (0.5 mg/ml) in a total volume of 160 ml. The pump is programmed to deliver 2-ml boluses at 6 to 8-minute lockout intervals with a background infusion rate at 1 ml/h. Patient-controlled analgesia is provided for at least 24 hours after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Patient-controlled analgesia is provided for at least 24 hours but no more than 48 hours. The pump is established with morphine (0.5 mg/ml) and dexmedetomidine (1.25 microgram/ml), in a total volume of 160 ml normal saline, and programmed to deliver 2-ml boluses at 6 to 8-minute lockout intervals with a background infusion rate of 1 ml/h.
  Other Names: Dexmedetomidine hydrochloride
  Arms: Dexmedetomidine group
Drug: Placebo — Patient-controlled analgesia is provided for at least 24 hours but no more than 48 hours. The pump is established with morphine (0.5 mg/ml), in a total volume of 160 ml normal saline, and programmed to deliver 2-ml boluses at 6 to 8-minute lockout intervals with a background infusion rate of 1 ml/h.
  Other Names: Normal saline
  Arms: Placebo group

SUMMARY:
Obstructive sleep apnea (OSA) is a common sleep disturbance that can cause intermittent hypoxia, hypercapnia, and sleep structure disorders. The presence of OSA is associated with worse outcomes after surgery including increased incidence of complications. High-flow nasal cannula (HFNC) therapy can improve oxygenation of OSA patients by maintaining a certain positive pressure in the nasopharyngeal cavity. Previous studies showed that, dexmedetomidine supplemented analgesia can improve sleep quality and pain relief. The investigators hypothesize that, for high-risk OSA patients following major non-cardiac surgery with HFNC therapy, dexmedetomidine supplemented analgesia can improve sleep quality. The purpose of this pilot randomized controlled trial is to investigate the impact of dexmedetomidine supplemented analgesia on sleep quality in high-risk OSA patients after major non-cardiac surgery.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common sleep disturbance that can cause intermittent hypoxia, hypercapnia, and sleep structure disorders; the latter include prolonged sleep latency, shortened sleep duration, frequent wake-up, and disordered circadian rhythm. During the postoperative period, surgical stress, pain and the residual effects of sedatives/analgesics can aggravate the sleep disorder and physiological changes in OSA patients. The resulting consequence is increased incidence of postoperative complications.

High-flow nasal cannula (HFNC) therapy can improve the oxygenation of OSA patients by forming a certain positive pressure in the nasopharyngeal cavity. Previous studies showed that HFNC therapy can reduce respiratory events, improve oxygenation in patients with moderate to severe OSA.

Dexmedetomidine is a highly selective α2-adrenoceptor agonist with sedative, analgesic and anti-anxiety properties. Unlike other sedative agents, dexmedetomidine exerts its sedative effects through an endogenous sleep-promoting pathway, producing a state like non-rapid eye movement sleep without disturbing respiration. Our previous studies shows that dexmedetomidine supplemented analgesia can improve sleep quality and pain relief in patients after surgery.

The investigators hypothesize that, for patients at high-risk of OSA who are recovering from major non-cardiac surgery and receiving HFNC therapy, dexmedetomidine supplemented analgesia can improve sleep quality and postoperative recovery. The purpose of this pilot randomized controlled trial is to investigate the impact of dexmedetomidine supplemented analgesia on the sleep quality in high-risk OSA patients after major non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years but <=80 years;
2. At high-risk of obstructive sleep apnea (a STOP-Bang score ≥3 combined with a serum bicarbonate ≥28 mmol/ L), but does not regularly receive continuous positive airway pressure (CPAP) therapy;
3. Scheduled to undergo major noncardiac surgery under general anesthesia, with an expected duration of >=1 hours and planned to use patient-controlled intravenous analgesia (PCIA) after surgery.

Exclusion Criteria:

1. Diagnosed as central sleep apnea syndrome;
2. Preoperative history of severe central nervous system diseases (epilepsy, parkinsonism, intracranial tumor, craniocerebral trauma) or neuromuscular disorders (myasthenia gravis);
3. History of schizophrenia or other mental disorders, or antidepressant or anxiolytic therapy within 3 month before surgery;
4. Inability to communicate in the preoperative period because of coma, profound dementia, deafness or language barriers;
5. History of drug or alcohol dependence, or sedative or hypnotic therapy within 1 month before surgery;
6. Contraindications to HFNC therapy (e.g. mediastinal emphysema, shock, cerebrospinal fluid leakage, nasosinusitis, otitis media, glaucoma);
7. Severe tracheal or pulmonary disease (e.g. bullous lung disease, pneumothorax, tracheal fistula);
8. Sick sinus syndrome, severe sinus bradycardia (<50 beats per minute), or second-degree or above atrioventricular block without pacemaker；
9. Severe hepatic dysfunction (Child-Pugh class C); Severe renal dysfunction (requirement of renal replacement therapy); severe heart dysfunction (preoperative New York Heart Association functional classification ≥3 or left ventricular ejection fraction <30%); ASA classification IV or above; or expected survival <24 hours after surgery;
10. Preoperative use of CPAP or HFNC therapy;
11. Expected intensive care unit (ICU) admission with tracheal intubation after surgery;
12. Refuse to participate in this study;
13. Other conditions that are considered unsuitable for study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
The percentage of non-rapid eye movement stage 2 (N2) sleep. | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Calculated according to polysomnographic monitoring results.

SECONDARY OUTCOMES:
Total sleep duration. | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Calculated according to polysomnographic monitoring results.
Sleep efficiency. | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  The ratio between the total sleep time and the total recording time and expressed as percentage. Calculated according to polysomnographic monitoring results.
Duration of non-rapid eye movement stage 1 (N1) sleep. | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Calculated according to polysomnographic monitoring results.
Percentage of non-rapid eye movement stage 1 (N1) sleep. | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Calculated according to polysomnographic monitoring results.
Duration of non-rapid eye movement stage 2 (N2) sleep. | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Calculated according to polysomnographic monitoring results.
Duration of non-rapid eye movement stage 3 (N3) sleep. | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Calculated according to polysomnographic monitoring results.
Percentage of non-rapid eye movement stage 3 (N3) sleep. | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Calculated according to polysomnographic monitoring results.
Duration of rapid eye movement sleep. | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Calculated according to polysomnographic monitoring results.
Percentage of rapid eye movement sleep. | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  Calculated according to polysomnographic monitoring results.
Sleep fragmentation index. | During the night of surgery (from 9 pm on the day of surgery to 6 am on the first day after surgery)
  The average number of arousals and awakenings per hour of sleep. Calculated according to polysomnographic monitoring results.

OTHER OUTCOMES:
Sedation level | Up to 5 days after surgery.
  Sedation level is assessed with the Richmond Agitation Sedation Scale (RASS), with scores ranging from -5 (unarousable) to +4 (combative) and 0 indicates alert and calm.
Cumulative morphine consumption | Up to 5 days after surgery.
  Cumulative morphine consumption
Pain intensity | Up to 5 days after surgery.
  Pain intensity is assessed twice daily (8-10 am and 18-20 pm) with the numeric rating scale, an 11-point scale where 0=no pain and 10=the worst pain.
Subjective sleep quality during the first 5 days after surgery. | Up to the fifth day after surgery.
  Subjective sleep quality is assessed daily (8-10 am) with the Richards-Campbell Sleep Questionnaire; which assesses subjective sleep quality in 5 aspects, each scale ranges from 0 to 100, with higher score indicating better function.
Incidence of delirium during the first 5 days after surgery. | Up to the fifth day after surgery.
  Delirium is assessed twice daily (8-10 am and 18-20 pm) with the 3D-Confusion Assessment Method for non-intubated patients or the Confusion Assessment Methods for the Intensive Care Unit for intubated patients.
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Incidence of postoperative complications within 30 days | Up to 30 days after surgery
  Postoperative complications are generally defined as newly occurred medical conditions that are deemed harmful and required therapeutic intervention within 30 days after surgery.
All-cause 30-day mortality | Up to 30 days after surgery
  All-cause 30-day mortality
Quality of life in 30-day survivors | At 30 days after surgery
  Quality of life is assessed with World Health Organization Quality of Life brief version (WHOQOL-BREF), a 24-item questionnaire that provides assessments of the quality of life in physical, psychological, social relationship, and environmental domains. For each domain, the score ranges from 0 to 100, with higher score indicating better function.
Cognitive function in 30-day survivors | At 30 days after surgery
  Cognitive function of 30-day survivors is assessed with the modified Telephone Interview for Cognitive Status (TICSm), a 12-item questionnaire that provides an assessment of global cognitive function by verbal communication via telephone. The score ranges from 0 to 48, with higher score indicating better function.
The overall subjective sleep quality in 30-day survivors | At 30 days after surgery
  Assessed with the Pittsburgh Sleep Quality Index, which estimates overall subjective sleep quality in the past 30 days. Overall score ranges from 0 to 21, with higher score indicating better sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Dong-Xin Wang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dempsey JA, Veasey SC, Morgan BJ, O'Donnell CP. Pathophysiology of sleep apnea. Physiol Rev. 2010 Jan;90(1):47-112. doi: 10.1152/physrev.00043.2008. PMID 20086074
- [Background] Benjafield AV, Ayas NT, Eastwood PR, Heinzer R, Ip MSM, Morrell MJ, Nunez CM, Patel SR, Penzel T, Pepin JL, Peppard PE, Sinha S, Tufik S, Valentine K, Malhotra A. Estimation of the global prevalence and burden of obstructive sleep apnoea: a literature-based analysis. Lancet Respir Med. 2019 Aug;7(8):687-698. doi: 10.1016/S2213-2600(19)30198-5. Epub 2019 Jul 9. PMID 31300334
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Background] Lee W, Nagubadi S, Kryger MH, Mokhlesi B. Epidemiology of Obstructive Sleep Apnea: a Population-based Perspective. Expert Rev Respir Med. 2008 Jun 1;2(3):349-364. doi: 10.1586/17476348.2.3.349. PMID 19690624
- [Background] Kapur VK, Auckley DH, Chowdhuri S, Kuhlmann DC, Mehra R, Ramar K, Harrod CG. Clinical Practice Guideline for Diagnostic Testing for Adult Obstructive Sleep Apnea: An American Academy of Sleep Medicine Clinical Practice Guideline. J Clin Sleep Med. 2017 Mar 15;13(3):479-504. doi: 10.5664/jcsm.6506. PMID 28162150
- [Background] Brown KA. Intermittent hypoxia and the practice of anesthesia. Anesthesiology. 2009 Apr;110(4):922-7. doi: 10.1097/ALN.0b013e31819c480a. PMID 19293703
- [Background] Fassbender P, Herbstreit F, Eikermann M, Teschler H, Peters J. Obstructive Sleep Apnea-a Perioperative Risk Factor. Dtsch Arztebl Int. 2016 Jul 11;113(27-28):463-9. doi: 10.3238/arztebl.2016.0463. PMID 27476705
- [Background] Kaw R, Pasupuleti V, Walker E, Ramaswamy A, Foldvary-Schafer N. Postoperative complications in patients with obstructive sleep apnea. Chest. 2012 Feb;141(2):436-441. doi: 10.1378/chest.11-0283. Epub 2011 Aug 25. PMID 21868464
- [Background] Hwang D, Shakir N, Limann B, Sison C, Kalra S, Shulman L, Souza Ade C, Greenberg H. Association of sleep-disordered breathing with postoperative complications. Chest. 2008 May;133(5):1128-34. doi: 10.1378/chest.07-1488. Epub 2008 Mar 13. PMID 18339794
- [Background] Liao P, Yegneswaran B, Vairavanathan S, Zilberman P, Chung F. Postoperative complications in patients with obstructive sleep apnea: a retrospective matched cohort study. Can J Anaesth. 2009 Nov;56(11):819-28. doi: 10.1007/s12630-009-9190-y. PMID 19774431
- [Background] Aloia MS, Stanchina M, Arnedt JT, Malhotra A, Millman RP. Treatment adherence and outcomes in flexible vs standard continuous positive airway pressure therapy. Chest. 2005 Jun;127(6):2085-93. doi: 10.1378/chest.127.6.2085. PMID 15947324
- [Background] Helviz Y, Einav S. A Systematic Review of the High-flow Nasal Cannula for Adult Patients. Crit Care. 2018 Mar 20;22(1):71. doi: 10.1186/s13054-018-1990-4. PMID 29558988
- [Background] McGinley BM, Patil SP, Kirkness JP, Smith PL, Schwartz AR, Schneider H. A nasal cannula can be used to treat obstructive sleep apnea. Am J Respir Crit Care Med. 2007 Jul 15;176(2):194-200. doi: 10.1164/rccm.200609-1336OC. Epub 2007 Mar 15. PMID 17363769
- [Background] Weerink MAS, Struys MMRF, Hannivoort LN, Barends CRM, Absalom AR, Colin P. Clinical Pharmacokinetics and Pharmacodynamics of Dexmedetomidine. Clin Pharmacokinet. 2017 Aug;56(8):893-913. doi: 10.1007/s40262-017-0507-7. PMID 28105598
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Zhang DF, Su X, Meng ZT, Li HL, Wang DX, Xue-Ying Li, Maze M, Ma D. Impact of Dexmedetomidine on Long-term Outcomes After Noncardiac Surgery in Elderly: 3-Year Follow-up of a Randomized Controlled Trial. Ann Surg. 2019 Aug;270(2):356-363. doi: 10.1097/SLA.0000000000002801. PMID 29742525
- [Background] Chung F, Abdullah HR, Liao P. STOP-Bang Questionnaire: A Practical Approach to Screen for Obstructive Sleep Apnea. Chest. 2016 Mar;149(3):631-8. doi: 10.1378/chest.15-0903. Epub 2016 Jan 12. PMID 26378880
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Katayama H, Kurokawa Y, Nakamura K, Ito H, Kanemitsu Y, Masuda N, Tsubosa Y, Satoh T, Yokomizo A, Fukuda H, Sasako M. Extended Clavien-Dindo classification of surgical complications: Japan Clinical Oncology Group postoperative complications criteria. Surg Today. 2016 Jun;46(6):668-85. doi: 10.1007/s00595-015-1236-x. Epub 2015 Aug 20. PMID 26289837
- [Derived] Sun P, Liang XQ, Chen NP, Ma JH, Zhang C, Shen YE, Zhu SN, Wang DX. Impact of mini-dose dexmedetomidine supplemented analgesia on sleep structure in patients at high risk of obstructive sleep apnea: a pilot trial. Front Neurosci. 2024 Oct 2;18:1426729. doi: 10.3389/fnins.2024.1426729. eCollection 2024. PMID 39416950